CLINICAL TRIAL: NCT06567028
Title: Prospective Evaluation of an OSPM-Enhanced Deep Learning Model for Identifying Premalignant and Malignant Ocular Surface Tumors
Brief Title: OSPM-Enhanced AI Model to Identify Premalignant and Malignant Ocular Surface Tumors
Status: Completed | Type: Observational
Sponsor: Ningbo Eye Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: NEH202408
Record Dates: First submitted 2024-08-20; First posted 2024-08-22 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Performance of the Model

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: OSPM-Enhanced AI Model — Analyze tumor images using the model developed in our study

SUMMARY:
An OSPM-enhanced deep learning model has been developed for identifying premalignant and malignant tumors using data retrospectively collected from the Ningbo Eye Hospital, Jiangdong Eye Hospital, and the Eye Hospital of Wenzhou Medical University. To further substantiate the model's effectiveness, we intend to evaluate it prospectively at Ningbo Eye Hospital.

ELIGIBILITY:
Inclusion Criteria:

● Ocular surface tumor images with histopathological findings

Exclusion Criteria:

● Low-quality images

Ages: 1 Year to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Child, Adult, Older Adult
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
AUROC | 3 months
  area under the receiver operating characteristic curve

CONTACTS AND LOCATIONS:
Locations (1):
- Ningbo Eye Hospital, Ningbo, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No